CLINICAL TRIAL: NCT03428594
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluation the Efficacy and Safety of Intravenous CKD-11101 Versus Darbepoetin Alfa in Patients Who Had Renal Anemia Receiving Hemodialysis
Brief Title: CKD-11101 Phase 3 IV Study in Patients Who Had Renal Anemia Receiving Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136Ane14004
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multi-center, phase 3 clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-11101 (Experimental): The dose of investigational product (Darbepoetin alfa) is adjusted according to the principles reflecting the MFDS (Ministry of Food and Drug Safety) approval for NESP, but is determined by the investigator's judgment considering various factors of the subjects that may affect the treatment of anemia.
  Interventions: Biological: CKD-11101
- NESP (Active Comparator): The dose of investigational product (Darbepoetin alfa) is adjusted according to the principles reflecting the MFDS (Ministry of Food and Drug Safety) approval for NESP, but is determined by the investigator's judgment considering various factors of the subjects that may affect the treatment of anemia.
  Interventions: Biological: NESP

INTERVENTIONS:
Biological: CKD-11101
  Arms: CKD-11101
Biological: NESP
  Arms: NESP

SUMMARY:
The aim of this study was to compare and evaluate efficacy and safety of intravenous CKD-11101 versus Darbepoetin alfa in patients who have renal anemia receiving hemodialysis.

DETAILED DESCRIPTION:
This study was designed as randomized, double-blind, multi-center, Phase 3 clinical study to evaluate the efficacy and safety of intravenous CKD-11101 versus Darbepoetin alfa in patients who had renal anemia receiving hemodialysis.

The selection criteria are evaluated for 19-year-old patients who receive stable hemodialysis treatment for 3 months or more in patients with chronic renal failure. After completion of the stabilization period of 12 to 16 weeks for Darbepoetin Alfa, the subjects with the mean Hb levels of 10 to 12g/dl measured during the baseline visit and 0 week visit are randomized to the test and control groups in a 1:1 ratio during the randomization visit. They have a 20-week maintenance period and a 4-week evaluation period.

ELIGIBILITY:
* Inclusion Criteria

  1. Patients with 19 years of age or older
  2. Patients with anemia in chronic renal failure
  3. Patients who started hemodialysis more than 3 months ago and receive appropriate hemodialysis, satisfying the following criterion:

     -Kt/V is ≥ 1.2 or Urea reduction ratio is ≥ 65%
  4. Patients with the mean Hb levels of 10 to 12g/dl measured at the baseline and randomization visits
  5. Patients with enough body iron stores who meet the following item:

     -Serum ferritin ≥ 100ng/ml or Transferrin saturation ≥ 20%
  6. Patients who have provided written consent to participate in the trial voluntarily
* Exclusion Criteria

  1. Patients with uncontrolled hypertension
  2. Patients who had hypersensitivity to erythropoietin agents
  3. Patients who had known hypersensitivity to mammalian cell-derived products or diluting agents
  4. Patients with history of severe cardiovascular diseases
  5. Patients who have received red blood cell transfusion or hormone therapy for anemia correction within 12 weeks prior to randomization
  6. Patients whose anemia is not caused by chronic renal failure or may affect anemia correction
  7. Patients whose AST/ALT test results performed at screening exceed twice of normal upper limit
  8. Patients who had experience of positive result in anti-erythropoietin antibody in previous treatment with erythropoiesis stimulating agent
  9. Patients who have been planned to change the dialysis method

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changed amount of mean hemoglobin level in evaluation period compared to the baseline | ([Mean of hemoglobin level measured in Weeks 20 - 24] - [Mean of hemoglobin level measured at Weeks -4 - 0])
  The equivalence test on mean hemoglobin level of test drug and to Reference Drug administration groups in evaluation period (Weeks 20 - 24) compared to the baseline (Weeks -4 - 0) will be conducted.
Mean administration dose in evaluation period: Mean dose administered in Weeks 20 - 24 | Weeks 20 - 24
  The equivalence test on mean administration dose of test drug and to Reference Drug administration groups in evaluation period (Weeks 20 - 24) will be conducted.

SECONDARY OUTCOMES:
Ratio of subjects who achieve target level of hemoglobin during the evaluation period | Weeks 20 - 24
  Ratio of subjects who maintain target level of hemoglobin: Compare the number of subjects who do not deviate from target level of hemoglobin during the evaluation period between groups
Mean hemoglobin levels at Weeks 20 and 24 | Weeks 20, 24
  Mean hemoglobin level at Weeks 20 and 24: Compare mean hemoglobin level at Weeks 20 and 24 between groups
Ratio of subjects who maintain hemoglobin level ≥ 10g/dl during maintenance period and evaluation period (interval of every 2 weeks) | Weeks 0 - 24
  Compare ratio of subjects who maintain hemoglobin level ≥ 10g/dl during maintenance period and evaluation period between groups (interval of every 2 weeks)
Ratio of subjects who changed dose during maintenance period and evaluation period | Weeks 0 - 24
  Ratio of subjects who changed dose: Compare ratio of subjects who change dose during maintenance period and evaluation period between groups
Ratio of subjects who receive transfusion during maintenance period and evaluation period | Weeks 0 - 24
  Ratio of subjects who receive red blood cell transfusion: Compare ratio of subjects who receive red blood cell transfusion during maintenance period and evaluation period between groups
Number of red blood cell transfusion per subject during maintenance period and evaluation period | Weeks 0 - 24
  Number of red blood cell transfusion per subject: Compare number of red blood cell transfusion per subject during maintenance period and evaluation period between groups

CONTACTS AND LOCATIONS:
Overall Officials: Su-Kil Park, M.D.,Ph.D., Principal Investigator — Asan Medical Center, College of Medicine, Univ. of Ulsan

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280